CLINICAL TRIAL: NCT02311127
Title: Comparing SecurAcath Versus StatLock to Secure Peripherally Inserted Central Catheters: a Randomised, Open Trial
Brief Title: SecurAcath Versus Statlock for PICC Securement
Acronym: SecurAstaP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S57358
Record Dates: First submitted 2014-11-28; First posted 2014-12-08 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-08

CONDITIONS: Patients With Any Condition Who Need a PICC for IV Therapy
Keywords: Peripherally Inserted Central Catheters; Securement device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SecurAcath (Experimental): Subcutaneous securement
  Interventions: Device: SecurAcath
- StatLock (Active Comparator): Adhesive securement
  Interventions: Device: StatLock

INTERVENTIONS:
Device: SecurAcath — Devices secures PICC subcutaneously and remains in place during the complete dwell time of the PICC
  Other Names: Subcutaneous catheter securement system
  Arms: SecurAcath
Device: StatLock — Device secures PICC however, device has to be changed weekly
  Other Names: Sutureless adhesive-backed device
  Arms: StatLock

SUMMARY:
Peripherally inserted central catheters (PICCs ) are used for the administration of intravenous fluids and for blood sampling. PICCs may remain in place for weeks to months and are safeguarded from migration or accidental dislodgement by securement devices. Different types of these devices are available. StatLock® (C.R. Bard) is a stabilization device with an adhesive anchor pad. The catheter wings of the PICC must be placed over the posts then the system is closed with "gull-wings" . StatLock® has to be changed weekly. Healthcare providers have to pay attention to prevent accidental catheter dislodgement during the renewal procedure. SecurAcath® (Interrad Medical) is a new securement device to the European market. The device uses a small subcutaneous anchor to secure the PICC. One of the advantages compared to adhesive stabilization devices, is a reduction in maintenance time by simplifying dressing changes and subsequently staff time. It is described that nurses report that care is left undone due to low staffing levels. Therefore, investigation of nursing time savings with the support of technology is imperative. SecurAcath® remains in place for life of the PICC and therefore has the potential to reduce the time for dressing change as there is no need for weekly device change. The objective of this study is to measure nursing time for dressing change and explore inserting and removal issues and patient experiences.

ELIGIBILITY:
Inclusion Criteria:

* Polyurethane PICC insertion
* Dutch speaking patient, able to give informed consent
* Intravenous treatment is administered in the University Hospitals Leuven

Exclusion Criteria:

* patients with known allergy to nickel or ethylene oxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time needed for dressing change | weekly during dressing change until catheter removal which is expected on an average after 2 weeks or up to 26 weeks

SECONDARY OUTCOMES:
Number of accidental removals | at catheter removal which is expected on an average after 2 weeks or up to 26 weeks
Number of catheters that migrated | weekly during dressing change until catheter removal which is expected on an average after 2 weeks or up to 26 weeks
  external catheter part will be measured
Catheter-related infection | at catheter removal which is expected on an average after 2 weeks or up to 26 weeks
  Labo confirmed catheter-related infection
Pain at catheter entry site related to device | every week with the catheter dressing change until catheter removal which is expected on an average after 2 weeks or up to 26 weeks
  measured by the VAS from 0 (no pain) to 10 (worst imaginable pain)
Ease of use of the device | at placement (day 1) and at catheter removal which is expected on an average after 2 weeks
  measured by the sumscore of the answers on 4 statements scored on a 5-item likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Godelieve A Goossens, PhD, RN, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Egan GM, Siskin GP, Weinmann R 4th, Galloway MM. A prospective postmarket study to evaluate the safety and efficacy of a new peripherally inserted central catheter stabilization system. J Infus Nurs. 2013 May-Jun;36(3):181-8. doi: 10.1097/NAN.0b013e3182893690. PMID 23558917
- [Background] Elen Hughes M. Reducing PICC migrations and improving patient outcomes. Br J Nurs. 2014 Jan 23-Feb 12;23(2):S12, S14-8. doi: 10.12968/bjon.2014.23.sup1.s12. PMID 24464053
- [Background] Alekseyev S, Byrne M, Carpenter A, Franker C, Kidd C, Hulton L. Prolonging the life of a patient's IV: an integrative review of intravenous securement devices. Medsurg Nurs. 2012 Sep-Oct;21(5):285-92. PMID 23243786
- [Derived] Goossens GA, Grumiaux N, Janssens C, Jerome M, Fieuws S, Moons P, Stas M, Maleux G. SecurAstaP trial: securement with SecurAcath versus StatLock for peripherally inserted central catheters, a randomised open trial. BMJ Open. 2018 Feb 24;8(2):e016058. doi: 10.1136/bmjopen-2017-016058. PMID 29478011